CLINICAL TRIAL: NCT02502708
Title: A Phase I Trial of Indoximod and Temozolomide-Based Therapy for Children With Progressive Primary Brain Tumors
Brief Title: Study of the IDO Pathway Inhibitor, Indoximod, and Temozolomide for Pediatric Patients With Progressive Primary Malignant Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG2105
Record Dates: First submitted 2015-07-06; First posted 2015-07-20 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Glioblastoma Multiforme; Glioma; Gliosarcoma; Malignant Brain Tumor; Ependymoma; Medulloblastoma; Diffuse Intrinsic Pontine Glioma; Primary CNS Tumor
Keywords: glioblastoma multiforme; glioma; gliosarcoma; malignant brain tumor; ependymoma; medulloblastoma
MeSH Terms: conditions — Glioblastoma; Glioma; Gliosarcoma; Brain Neoplasms; Ependymoma; Medulloblastoma; Diffuse Intrinsic Pontine Glioma | interventions — 1-methyltryptophan; Temozolomide; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (CLOSED) (Experimental): Core Regimen: Dose-escalation of indoximod, in combination with temozolomide, for pediatric patients with progressive brain tumors.
  Indoximod will be administered in escalating doses. Initial dosing will be 12.8 mg/kg/dose BID with escalation planned to 22.4 mg/kg/dose BID.
  Temozolomide to be given at 200 mg/m^2 x 5 days
  Interventions: Drug: Indoximod; Drug: Temozolomide
- Group 2 (CLOSED) (Experimental): Expansion cohorts: Indoximod therapy at the pediatric recommended phase 2 dose (RP2D) determined by Group 1, in combination with temozolomide.
  Indoximod will be administered at the RP2D of 19.2 mg/kg/dose BID.
  Temozolomide to be given at 200 mg/m^2 x 5 days
  Interventions: Drug: Indoximod; Drug: Temozolomide
- Group 3 (CLOSED) (Experimental): Dose-escalation of indoximod, in combination with up-front conformal radiation therapy, for pediatric patients with progressive brain tumors.
  Indoximod will be administered in escalating doses. Initial dosing will be 12.8 mg/kg/dose BID with escalation planned to 22.4 mg/kg/dose BID.
  Temozolomide to be given at 200 mg/m^2 x 5 days
  Interventions: Drug: Indoximod; Drug: Temozolomide; Radiation: Conformal Radiation
- Group 3b (Experimental): Indoximod, in combination with up-front conformal radiation therapy, for pediatric patients with newly diagnosed treatment-naive diffuse intrinsic pontine glioma (DIPG).
  Indoximod will be administered at the RP2D of 19.2 mg/kg/dose BID.
  Temozolomide to be given at 200 mg/m^2 x 5 days
  Interventions: Drug: Indoximod; Drug: Temozolomide; Radiation: Conformal Radiation
- Group 4 (Experimental): Continued access to indoximod in combination with low-dose oral cyclophosphamide and etoposide for patients with progressive disease after treatment with indoximod plus temozolomide.
  Indoximod will be administered at 32 mg/kg/dose divided twice daily.
  Cyclophosphamide to be given at 2.5 mg/kg/dose daily
  Etoposide to be given at 50 mg/m2/dose daily
  Interventions: Drug: Indoximod; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Indoximod — Indoximod will be administered orally twice daily.
  Other Names: 1-methyl-D-tryptophan; D-1MT
Drug: Temozolomide — Temozolomide will be administered on days 1-5 of every 28 day cycle.
  Other Names: Temodar; Methazolastone
  Arms: Group 1 (CLOSED); Group 2 (CLOSED); Group 3 (CLOSED); Group 3b
Radiation: Conformal Radiation — Conformal radiation will be administered on days 3-7 of induction cycle.
  Arms: Group 3 (CLOSED); Group 3b
Drug: Cyclophosphamide — Cyclophosphamide will be administered orally daily.
  Arms: Group 4
Drug: Etoposide — Etoposide will be administered orally daily.
  Arms: Group 4

SUMMARY:
This is a first-in-children phase 1 trial using indoximod, an inhibitor of the immune "checkpoint" pathway indoleamine 2,3-dioxygenase (IDO), in combination with temozolomide-based therapy to treat pediatric brain tumors. Using a preclinical glioblastoma model, it was recently shown that adding IDO-blocking drugs to temozolomide plus radiation significantly enhanced survival by driving a vigorous, tumordirected inflammatory response. This data provided the rationale for the companion adult phase 1 trial using indoximod (IND#120813) plus temozolomide to treat adults with glioblastoma, which is currently open (NCT02052648). The goal of this pediatric study is to bring IDO-based immunotherapy into the clinic for children with brain tumors. This study will provide a foundation for future pediatric trials testing indoximod combined with radiation and temozolomide in the up-front setting for patients with newly diagnosed central nervous system tumors.

ELIGIBILITY:
Eligibility Criteria

* Age: 3-21 years.
* Group 1 or Group 3: histologically proven initial diagnosis of primary malignant brain tumor, with no known curative treatment options.
* Group 2: histologically proven initial diagnosis of high-grade glioma (WHO grade III and IV), ependymoma, medulloblastoma, or other primary central nervous system tumor.
* Group 3b: Patients with a radiographic diagnosis or histologically proven diagnosis of diffuse intrinsic pontine glioma (DIPG).
* MRI confirmation of tumor progression or regrowth.
* Patients must be able to swallow whole capsules.
* Patients with metastatic disease are eligible for enrollment.
* Lansky or Karnofsky performance status score must be > 50%.
* Seizure disorders must be well controlled on antiepileptic medication.
* DIPG patients enrolled to Group 3b must not have been previously treated with radiation or any medical therapy.
* Patients previously treated with temozolomide, cyclophosphamide, and/or etoposide are eligible for enrollment.

Exclusion Criteria

* Prior invasive malignancy, other than the primary central nervous system tumor, unless the patient has been disease free and off therapy for that disease for a minimum of 3 years
* Patients with baseline QTc interval of more than 470 msec at study entry, and patients with congenital long QTc syndrome.
* Active autoimmune disease

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2015-10; Primary Completion 2019-12-12 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of regimen limiting toxicities (RLTs) | First 28 days of treatment
  To estimate the RP2D of indoximod combined with temozolomide
Objective Response Rate | Up to three years
  To assess preliminary evidence of efficacy of indoximod and temozolomide using COG brain tumor measurement criteria.
Incidence of regimen limiting toxicities (RLTs) | First 35 days of treatment
  To estimate the RP2D of indoximod combined with conformal radiation
Safety and tolerability assessed by development of AEs and laboratory parameters of indoximod in combination with cyclophosphamide and etoposide. | Up to three years
  In patients who initially achieve prolonged stable disease or better with Indoximod plus temozolomide but then develop progressive disease

SECONDARY OUTCOMES:
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | First 48 hours of treatment
  Group 1
Safety and Tolerability of Indoximod combined with Temozolomide as assessed by incidence and severity of adverse events, dose interruptions and dose reductions. | Continuous during study until 30 days after study treatment is complete.
  Group 1 and 2
Progression Free Survival (PFS) | Up to three years
  Group 2
Time to Progression | Start of study until disease progression follow-up, up to three years
  Group 2
Overall Survival | Start of study until end of follow-up, up to five years
  Group 2
Safety and Feasibility of Indoximod combined with conformal radiation as assessed by incidence and severity of adverse events, dose interruptions and dose reductions. | Continuous during study until 30 days after study treatment is complete.
  Group 3

CONTACTS AND LOCATIONS:
Overall Officials: Gene Kennedy, MD, Study Director — NewLink Genetics Corporation
Locations (5):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Children's Heathcare of Atlanta, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Johnson TS, MacDonald TJ, Pacholczyk R, Aguilera D, Al-Basheer A, Bajaj M, Bandopadhayay P, Berrong Z, Bouffet E, Castellino RC, Dorris K, Eaton BR, Esiashvili N, Fangusaro JR, Foreman N, Fridlyand D, Giller C, Heger IM, Huang C, Kadom N, Kennedy EP, Manoharan N, Martin W, McDonough C, Parker RS, Ramaswamy V, Ring E, Rojiani A, Sadek RF, Satpathy S, Schniederjan M, Smith A, Smith C, Thomas BE, Vaizer R, Yeo KK, Bhasin MK, Munn DH. Indoximod-based chemo-immunotherapy for pediatric brain tumors: A first-in-children phase I trial. Neuro Oncol. 2024 Feb 2;26(2):348-361. doi: 10.1093/neuonc/noad174. PMID 37715730